CLINICAL TRIAL: NCT05502666
Title: ¡Salud! Por la Vida: A Colorectal Screening Promotion Program for Patients Attending Federally Qualified Health Centers in Puerto Rico.
Brief Title: ¡Salud! Por la Vida (SPLV) A Colorectal Screening Promotion Program
Acronym: SPLV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); M.D. Anderson Cancer Center (Other); National Cancer Institute (NCI) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Vivian Colon, Professor, University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A8060116
Record Dates: First submitted 2022-08-04; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer
Keywords: Hispanic/Latino; Behavioral Intervention; Lay Health Workers; Colorectal cancer; Colorectal cancer screening; Colonoscopy; cancer prevention
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Intervention Arm: ¡Salud! Por la vida Educational Intervention After completing eligibility and baseline surveys, trained lay health workers delivered an educational intervention for colorectal cancer screening with included a tailored interactive multimedia intervention (TIMI), newsletter, infographics, and a provider prompt for colorectal cancer screening. This educational session was delivered at intervention clinics and lasted about 1 hour. Follow-up data was collected starting at 6 months post educational session.
  Interventions: Behavioral: ¡Salud! Por la Vida
- Control Arm (No Intervention): Control Arm: No intervention was delivered. At baseline, participants completed eligibility and baseline surveys. Follow-up data was collected 6 months post-baseline survey.

INTERVENTIONS:
Behavioral: ¡Salud! Por la Vida — Lay health worker (LHW) delivered educational intervention for colorectal cancer screening (CRCS). The intervention consisted in having the participant complete a tailored interactive multimedia intervention (TIMI). TIMI consisted of a series of educational videos that addressed common barriers to colorectal cancer screening as well as provided information about colorectal cancer (CRC) and CRCS tests. Participants were able to tailor the TIMI for sex (male/female) and CRC family history. After TIMI completion, the LHW provided participant with a copy of the SPLV newsletter and printed infographics on CRC, CRCS, and an action plan tailored by type of CRCS (FOBT/FIT or colonoscopy). The Intervention Group subject participation took approx. up to 2 hours and Control Group up to 1 hour (half hour for each: baseline and follow-up interview). Follow-up data was collected 6 months post education session (intervention group) or post-baseline survey (control group).
  Arms: Intervention Arm

SUMMARY:
The overall goal of this educational program was to increase colorectal cancer screening (CRCS) in men and women who attend Federally Qualified Health Centers (FQHC) in Puerto Rico. FQHCs, referred to in Puerto Rico as "Clínicas 330", are ideal settings to implement innovative approaches to increase CRCS because they serve primarily low-income patients who typically have lower rates of screening. The goal of this study, is to develop and evaluate the impact of a clinic level intervention on increasing CRCS among low-income Puerto Rican men and women aged 50-75, who have either never been screened for colorectal cancer, or are under-screened according recommended guidelines. To evaluate the delivery of the CRCS education program we used a group randomized controlled trial that provided data to determine the effectiveness of the CRC intervention program compared with usual practice (no intervention).

ELIGIBILITY:
Inclusion Criteria:

* Female aged 50-75, patient at a participating FQHC.
* Male aged 50-75, patient at a participating FQHC.

Exclusion Criteria:

* Having completed a fecal occult blood test (FOBT) or a fecal immunochemical test (FIT) in the past year.
* Having completed a sigmoidoscopy in the last 5 years.
* Having completed a colonoscopy in the last 10 years.
* Prior history of colorectal cancer.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2017-07-08 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Colorectal Cancer Screening | 6 months after the intervention
  Number of participants aged 50-75 who completed a colorectal cancer screening (FOBT, FIT, and/or colonoscopy) Screening behavior status at follow-up was assessed by asking patients the month and year of their last CRCS and by medical record review.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Puerto Rico, Medical Sciences Campus, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serra YA, Colon-Lopez V, Savas LS, Vernon SW, Fernandez-Espada N, Velez C, Ayala A, Fernandez ME. Using Intervention Mapping to Develop Health Education Components to Increase Colorectal Cancer Screening in Puerto Rico. Front Public Health. 2017 Dec 7;5:324. doi: 10.3389/fpubh.2017.00324. eCollection 2017. PMID 29270400
- [Background] Colon-Lopez V, Valencia-Torres IM, Rios EI, Llavona J, Velez-Alamo C, Fernandez ME. Knowledge, Attitudes, and Beliefs About Colorectal Cancer Screening in Puerto Rico. J Cancer Educ. 2023 Apr;38(2):552-561. doi: 10.1007/s13187-022-02153-z. Epub 2022 Mar 31. PMID 35359256
- See also: ¡Salud! por la Vida Educational Materials in Spanish — https://canceroutreachpr.org/salud-por-la-vida/
- See also: ¡Salud! por la Vida Educational Materials in English — https://sph.uth.edu/research/centers/chppr/research/puerto-rico/index.htm